CLINICAL TRIAL: NCT06657534
Title: SISIPUSH: Evaluation of Hemolysis and Iatrogenic Anemia Using the Push-pull Method to Obtain Blood from Pediatric Patients with Central Venous Catheters
Acronym: SISIPUSH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ONZ-2024-0215
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Pediatrics; Central Venous Catheter
Keywords: push-pull technique
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Push-pull technique
  Interventions: Procedure: Push-pull technique
- Control (Active Comparator): Standard of care blood sampling method with waste blood
  Interventions: Procedure: SOC (Standard of care)

INTERVENTIONS:
Procedure: Push-pull technique — push-pull technique as described by McBride et al, J Infus Nurs 2018
  Arms: Intervention
Procedure: SOC (Standard of care) — Standard of care method to obtain blood with waste blood
  Arms: Control

SUMMARY:
Anemia is frequently observed during hospitalizations, both in adults and children. In addition to the fact that anemia can be caused by an acute or chronic condition, blood samples taken during the hospital stay contribute to additional blood loss (so-called iatrogenic anemia).

For children, the relative amount of blood taken at each blood collection is greater than in adults. It is therefore expected that in children, due to the lower circulating blood volume, the relative impact of repeated blood sampling is greater and interventions such as sparing the number of blood samples or blood volume can have a relevant impact on the onset of anemia, the need for iron supplements or blood transfusions and the general clinical recovery.

For children, only limited data are available on the development of iatrogenic anemia during hospital stay. In a study of children in an intensive care unit, a decrease in hemoglobin of 0.7 g/dl can already be seen with an average stay of 4.5 days (and an average number of blood samples of 2.9) (François et al. Ped Crit Car Med, 2022). The average blood volume lost to blood samples during the stay is 3.9 ml/kg, which already corresponds to 5% of the total blood volume. Interventions to decrease the frequency of blood sampling or to perform the same analyses on a smaller blood volume (e.g. adapted, smaller blood tubes for children) are therefore useful in preventing the development of anemia during a hospital stay, especially in children.

Alternative methods have been described to save on blood volume when performing blood sampling, especially if these are performed via central venous catheters (surgically or non-surgically placed). To obtain a suitable sample via such catheters, the usual technique is to obtain 5 to 10 ml of blood and discard the volume (so-called "waste blood") before the sample for laboratory analysis is obtained (typically only 1-2 ml). A recently published technique is the so-called push-pull method (described by McBride et al, J Infus Nurs 2018), in which blood sampling can be performed without waste blood.

The push-pull technique has been studied in children, but mainly in oncological and intensive care units. Paired analyses have verified that the technique provides a reliable sample for most blood analyses, including blood count, electrolytes, liver and kidney function parameters, CRP, but also coagulation factors and therapeutic drug monitoring. The occurrence of complications, of which the development of catheter-related bacteremia is of particular importance, is not described. A beneficial effect on anemia onset has not yet been described, usually due to low patient numbers per study (23-35 patients).

In SISIPUSH, we compare the push-pull technique with the standard-of-care in hospitalised children who undergo blood sampling via a central venous catheter for diagnostic reasons (in the context of routine care). By means of a 1:1 randomization, eligible patients who gave informed consent are assigned to one of the two methods for the remainder of the hospitalization. From the moment of randomization until discharge from the hospital, data will be collected from the medical file that are collected routinely (number of blood samples, hemoglobin values, number of blood transfusions, markers of hemolysis, age and gender, reason for hospitalization, type of catheter) and compared between the two groups. In parallel, nurses score the easy of use and satisfaction with the procedure at each blood sample.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patient at the Specialist Pediatric Department of Ghent University Hospital
* age 0-18 years
* presence of a central venous catheter for diagnostic or therapeutic reasons of the type surgically placed (Hickman, port-a-cath) or non-surgically placed (vena jugularis interna, subclavia, femoralis,...)
* patent catheter with possibility of infusion of fluids and collection of blood on at least one of the lumens
* clinical and/or radiographic confirmation of correct central position of the catheter tip
* at least one blood collection per week hospitalization expected or already planned

Exclusion Criteria:

* presence of a bloodstream or catheter related infection before or at the time of randomization

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of hemoglobin | from randomization to discharge from the hospital or removal of the central venous catheter
  trend of hemoglobin (from the first blood draw after randomization to the last blood draw during the same hospitalization), which is defined as the sum of the negative differences of hemoglobin determinations (grams per deciliter) between two consecutive blood draws

SECONDARY OUTCOMES:
Hemolysis | from randomization to discharge from the hospital or removal of the central venous catheter
  analysis of hemolysis parameters on all blood samples (distribution of serum potassium and lactate dehydrogenase between the two study populations)
Anemia onset | from randomization to discharge from the hospital or removal of the central venous catheter
  proportion of patients diagnosed with anemia (hemoglobin <7 g/dl) during hospitalization
Need for erytrocyte transfusion | from randomization to discharge from the hospital or removal of the central venous catheter
  number of patients undergoing a packed red blood cell transfusion during hospitalization, expressed as proportion of patients compared to total number of patients, in number of transfusions per total number of blood samples and in number of transfusions per day of hospitalization since inclusion
Hemolytic samples | from randomization to discharge from the hospital or removal of the central venous catheter
  proportion of blood samples reported by the clinical laboratory as hemolytic
Failed blood samples | from randomization to discharge from the hospital or removal of the central venous catheter
  proportion of blood samples that were not analyzable and reason for this (hemolysis or other)
Bacteremia onset | from randomization to discharge from the hospital or removal of the central venous catheter
  proportion of patients with bacteremia (positive blood culture) during the course of the study
Catheter dysfunction | from randomization to discharge from the hospital or removal of the central venous catheter
  proportion of patients in whom the central venous catheter had to be removed early due to dysfunction or infection
Operator ease of use | from randomization to discharge from the hospital or removal of the central venous catheter
  assessment of satisfaction (0-5) and complexity (0-5) of the procedure by the healthcare personnel performing the blood sampling

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
peer-reviewed publication
Supporting Information: Study Protocol, CSR
Time Frame: January 2026